CLINICAL TRIAL: NCT03966677
Title: Sensory Abnormalities in Post-surgical Peripheral Neuropathy: A Comparison of Subjects With and Without Severe Pain Using Normative Data
Brief Title: Sensory Abnormalities in Post-surgical Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, mads u werner, Principal Investigator, University of Copenhagen
Other Study IDs: H-16034340
Record Dates: First submitted 2019-05-25; First posted 2019-05-29 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain
Keywords: Groin hernia repair; Persistent postsurgical pain; Quantitative sensory testing (QST); Normative data
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- P-GHR: Patients with persistent severe pain after groin hernia repair.
- NP-GHR: Patients without pain after groin hernia repair.
- NP: Healthy non-operated controls

SUMMARY:
The concept of normality is a cornerstone in medical practice and research. As an example, in clinical chemistry, a laboratory value based on a plasma sample exceeding the +/- 1.96 x standard deviation (SD) range, referenced from normative material, is, per definition, outside the normal range (the reference interval). Obviously, a number of reasons for this deviation may exist. The sample value could reflect a "true" pathological condition but could also be caused by error, e.g., technical measurement error, drug-interaction error, random error, or reflect a value occurring in 5% of the healthy population. Conversely, a sample value in the normal range evidently does not exclude a pathological condition.

The reference interval is calculated from a large number of healthy subjects sampled across age, anthropometrics, ethnicity, and gender. Normative reference intervals are certainly of help, particularly in the screening of subjects, but may be of limited value in the detailed assessment of pathophysiological processes. Also, increasing the number of analyses in a subject expands the risk of making a type I error (acquiring "false" positive results). The likelihood of one or more type I errors in the analysis of 10 different laboratory values in one subject is impressive 46% ([1 - 0.95^10] =0.46). It is well-known that multiple measurements are commonly performed in medical practice and research, but corrected significance levels are not always used.

DETAILED DESCRIPTION:
Quantitative sensory testing (QST) is defined as perceptually quantifiable responses to graded chemical (capsaicin), electrical, mechanical (pressure, punctate, vibratory, and light touch), or thermal (cool, warmth, cold pain, and heat pain) stimuli. Thus, QST is a psychophysical method primarily assessing small nerve fiber function in the skin. The method is ubiquitously used for the assessment of peripheral neuropathies, e.g., chemotherapy-induced neuropathy, painful diabetic polyneuropathy, post-herpetic neuralgia, and post-surgical neuropathy. Sensory mapping and QST are essential tools in grading definite or probable neuropathic pain, as stated in the definition: "Demonstration of the distinct neuroanatomically plausible distribution by at least one confirmatory test." Thus, examining somatosensory profiles in chronic post-surgical pain (CPSP) could be an important step in distinguishing the pathophysiologic components behind the transition from acute to chronic pain. However, determining when a measured variable is abnormal is obviously of prime importance in somatosensory research. During the last decade, the German Research Network on Neuropathic Pain (DFNS) has acquired normative sensory data from healthy individuals using a standardized testing protocol. Clearly, a deviating sensory response from an individual with a painful peripheral neuropathy could be evaluated by use of these normative data and eventually be classified as an abnormal response (absolute approach).

However, other alternatives exist that, hypothetically, might provide improved diagnostic specificity and sensitivity. First, in unilateral sensory deficits (mono-neuropathies), assessments at the contralateral side are possible, allowing a comparison with the pathological side (relative approach). The within-subject variances (WSV) are often significantly smaller than the between-subject variances (BSV) in QST assessments. In a normative study including thermal assessments (n = 100), the WSV and the BSV ranged between 18-23% and 77-82% of the total variance, respectively. Correspondingly, in a study of individuals with post-thoracotomy pain syndrome, the estimated WSV and BSV were 5-28% and 72-95%, respectively. Thus, scenarios using the subject as their own control may reduce data variability and improve diagnostic efficacy. However, the use of a contralateral homologous area as a control area in sensory testing has been questioned by several authors. The occurrence of mirror image sensory dysfunction (MISD) may affect contralateral assessments, requiring a distant control area. Second, instead of using healthy controls in pain studies, the use of post-surgical pain-free individuals as controls (e.g. post-groin hernia repair, post-thoracotomy) has been recommended in chronic post-surgical pain studies.

In spite of the importance of selecting an optimally controlled research design, the research group is only aware of one QST study addressing the control-group problem, i.e., a study including individuals with complex regional pain syndrome type I (CRPS I) restricted to one extremity. The study examined the validity of using the contralateral side as a control compared to using normative data from healthy individuals. The study recommended that the contralateral side in CPRS I individuals should be used as a control (relative approach).

Thus, it may be inferred that the following approaches are available for evaluating sensory data from an anticipated pathological site: an empirical approach (á priori set reference values), an absolute approach (comparing the subject's pathological side with normative data), and a relative approach (comparing the subject's side-to-side differences with normative data).

The present study has a prospective, observational, three-cohort design comparing somatosensory profiles from a cohort with groin hernia repair (GHR) associated CPSP (P-GHR; n = 70) across two standard cohorts: one surgical cohort without CPSP (NP-GHR; n = 54) and another healthy non-surgical cohort (NOP; n = 54). Testing sites are the surgical groin, with the comparator sites, the non-surgical groin, and the lower arm. The QST assessments are compared across cohorts (P-GHR, NP-GHR, NOP), testing sides (surgical side, non-surgical side), and testing sites (groins, arm). The statistical processing is by linear mixed-effects models and z-transformations, using the NOP cohort as reference material.

The main objective is:

* To characterize and interpret the pathophysiologic substrate behind the somatosensory profiles in individuals with GHR-associated CPSP using relevant controls

Other objectives are:

* To examine the somatosensory data repeatability
* To determine the diagnostic efficiency of QST in identifying GHR-associated somatosensory abnormalities
* To compare the somatosensory testing efficacy of the absolute approach compared to the relative approach, using normative healthy controls
* To examine contralateral somatosensory abnormalities in individuals with/without GHR-associated CPSP

ELIGIBILITY:
INCLUSION CRITERIA:

All study subjects must meet all the following criteria to be eligible to enroll in the study:

* Age above 18 yrs and below 65 yrs
* Signed informed consent
* Body mass index (BMI): 18 < BMI < 35 kg/m^2
* ASA I-II

In addition, for study subjects without pain after GHR (NP-GHR):

* having undergone uncomplicated, elective, unilateral open GHR a.m. Lichtenstein
* no restriction in ADL-functions due to the GHR
* activity-related groin pain < 3 (numerical rating scale [NRS]: 0 = no pain, 10 = worst imaginable pain)

EXCLUSION CRITERIA:

Any study subject, who meets one or more of the following criteria, is not suitable for inclusion in this study:

* do not speak or understand Danish
* who cannot cooperate with the investigation
* abuse of alcohol or drugs - according to investigator's evaluation
* use of psychotropic drugs (exception of SSRI)
* neurologic or psychiatric disease
* chronic pain condition
* regular use of analgesic drugs
* skin lesions or tattoos in the assessment areas (groins, lower arm)
* nerve lesions in the assessment sites (e.g., after trauma, abdominal surgery)

In addition, for healthy non-operated study subjects (NP):

* subjects, who have had previous surgery in or near the groin region
* use of prescription drugs one week before the trial
* use of over-the-counter (OTC) drugs 48 hours before the trial
* experiencing pain at rest > 3 (NRS)
* experiencing activity-related pain in or near the groin > 3 (NRS)

In addition, for study subjects without pain after GHR (NP-GHR):

* experiencing pain at rest > 3 (NRS)
* experiencing activity-related pain in or near the groin > 3 (NRS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects with pain after GHR (P-GHR) (n=54) Study subjects without pain after GHR (NP-GHR) (n=54) Healthy non-operated study subjects (NP) (n=54)
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Thermal thresholds | 2019-2023
  Warmth detection threshold (WDT), cool detection threshold, heat pain threshold (HPT) and cold pain threshold (CPT) are made by a computerized contact thermode (Thermotest, Somedic AB, Sweden) with an active thermal surface of 12.5 cm^2 (2.5 x 5.0 cm^2) as previously described in detail. The thresholds are determined from a baseline temperature of 32°C with a ramp rate of + 1°C/s. Cut-offs for heat and cold are 50°C and 5°C, respectively. The assessments are made in triplicate and the mean values are used in the statistical analyses.
Pressure algometry | 2019-2023
  Deep-tissue pain sensitivity is assessed using a hand-held pressure algometer with a neoprene-coated tip of area 1.0 cm2 (Somedic AB, Sweden), as previously described. The algometer is applied perpendicularly to the skin with a pressure rate of 30 kPa/s. The study subject is told to report the pressure pain threshold (PPT) by activating the button device when pain is perceived. The cut-off limit is 350 kPa. Testing is done in triplicate and the average value is used in the statistical analyses.
Suprathreshold heat stimulation | 2019-2023
  A short tonic heat stimulus (heating area 12.5 cm^2; ramp rate: 1°C/s, plateau: 47°C, 5 s; STH) is delivered in order to evaluate the suprathreshold heat pain perception (NRS).
Sensory mapping | 2019-2023
  Sensory mapping in the groin areas is assessed with a 25°C metal roll (Somedic AB), moved at a rate of 1 to 2 cm/s from skin with normal cool perception, using an octagonal approach, into the areas in order to indicate sensory changes. Changes in the study subject's cool perception are indicated by a marker on the skin, and subsequently transferred to a transparent sheet for later area assessment in a vector-based drawing drawing program (Canvas 12.0; ACD Systems, Seattle, WA).
Tactile thresholds | 2019-2023
  Tactile detection thresholds (TDT) and tactile pain threshold (TPT) are determined by polyamide monofilaments (Stoelting, IL, USA; nominal buckling force ranging from 0.04 to 4,400 mN) using a modified Dixon up-and-down method, with 3 descending and 3 ascending stimulus intensities. The filament with the smallest buckling force leading to tactile recognition (TDT) is registered. The tactile pain threshold (TPT) is determined by the same stimulus paradigm, but registering the perception of pain (sharpness/sting; TPT).
Temporal summation | 2019-2023
  Temporal summation test, i.e., the perception in response to repetitive (0.3 to 3 Hz) mechanical stimulation [i.e., wind-up like pain: WUP], indicates presence of central sensitization. The repetitive 1 Hz stimuli for 60 s are either dynamically delivered by a brush or statically delivered by a polyamide filament (one nominal rank below TPT). The study subjects are told to report the level of pain (NRS) every 15 s-1 during the stimulation. Signs of aftersensations are followed 60 s after discontinuation of the stimulation, and the intensity of discomfort or pain is rated by NRS.

SECONDARY OUTCOMES:
Assessments of Anxiety and Depression | 2019-2023
  Hospital Anxiety and Depression Scale (HADS; 14 items scale; 0-21 units)
Assessment of Pain Catastrophizing | 2019-2023
  Pain Catastrophizing Scale (PCS; 13 item scale; 0-65 units)

CONTACTS AND LOCATIONS:
Locations (1):
- Multidisciplinary Pain Center 7612, Neuroscience Center, Rigshospitalet, Blegdamsvej 9, Copenhagen O, Denmark

IPD SHARING:
Plan to Share IPD: Yes
https://register.clinicaltrials.gov/prs/app/template/EditProtocol.vm?listmode=Edit&uid=U000190V&ts=15&sid=S0008RBK&cx=-gmj8tv
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Treede RD. The role of quantitative sensory testing in the prediction of chronic pain. Pain. 2019 May;160 Suppl 1:S66-S69. doi: 10.1097/j.pain.0000000000001544. PMID 31008852
- [Background] Reimer M, Forstenpointner J, Hartmann A, Otto JC, Vollert J, Gierthmuhlen J, Klein T, Hullemann P, Baron R. Sensory bedside testing: a simple stratification approach for sensory phenotyping. Pain Rep. 2020 May 21;5(3):e820. doi: 10.1097/PR9.0000000000000820. eCollection 2020 May-Jun. PMID 32903958
- [Background] Truini A, Aleksovska K, Anderson CC, Attal N, Baron R, Bennett DL, Bouhassira D, Cruccu G, Eisenberg E, Enax-Krumova E, Davis KD, Di Stefano G, Finnerup NB, Garcia-Larrea L, Hanafi I, Haroutounian S, Karlsson P, Rakusa M, Rice ASC, Sachau J, Smith BH, Sommer C, Tolle T, Valls-Sole J, Veluchamy A. Joint European Academy of Neurology-European Pain Federation-Neuropathic Pain Special Interest Group of the International Association for the Study of Pain guidelines on neuropathic pain assessment. Eur J Neurol. 2023 Aug;30(8):2177-2196. doi: 10.1111/ene.15831. Epub 2023 May 30. PMID 37253688
- [Background] Finnerup NB, Haroutounian S, Kamerman P, Baron R, Bennett DLH, Bouhassira D, Cruccu G, Freeman R, Hansson P, Nurmikko T, Raja SN, Rice ASC, Serra J, Smith BH, Treede RD, Jensen TS. Neuropathic pain: an updated grading system for research and clinical practice. Pain. 2016 Aug;157(8):1599-1606. doi: 10.1097/j.pain.0000000000000492. PMID 27115670
- [Background] Pfau DB, Krumova EK, Treede RD, Baron R, Toelle T, Birklein F, Eich W, Geber C, Gerhardt A, Weiss T, Magerl W, Maier C. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): reference data for the trunk and application in patients with chronic postherpetic neuralgia. Pain. 2014 May;155(5):1002-1015. doi: 10.1016/j.pain.2014.02.004. Epub 2014 Feb 10. PMID 24525274
- [Background] Magerl W, Krumova EK, Baron R, Tolle T, Treede RD, Maier C. Reference data for quantitative sensory testing (QST): refined stratification for age and a novel method for statistical comparison of group data. Pain. 2010 Dec;151(3):598-605. doi: 10.1016/j.pain.2010.07.026. Epub 2010 Oct 20. PMID 20965658
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Background] Kemler MA, Schouten HJ, Gracely RH. Diagnosing sensory abnormalities with either normal values or values from contralateral skin: comparison of two approaches in complex regional pain syndrome I. Anesthesiology. 2000 Sep;93(3):718-27. doi: 10.1097/00000542-200009000-00021. PMID 10969305
- [Background] Rosenberger DC, Pogatzki-Zahn EM. Chronic post-surgical pain - update on incidence, risk factors and preventive treatment options. BJA Educ. 2022 May;22(5):190-196. doi: 10.1016/j.bjae.2021.11.008. Epub 2022 Feb 24. No abstract available. PMID 35496645